CLINICAL TRIAL: NCT04794972
Title: An Open-Label, Multi-Center, Phase I Study to Evaluate the Safety, Tolerability，Pharmacokinetic/Pharmacodynamics and Anti-tumor Activity of Tetra-specific Antibody GNC-039 in Participants With Relapsed/Refractory or Metastatic Solid Tumors
Brief Title: A Study of GNC-039, a Tetra-specific Antibody, in Participants With Relapsed/Refractory or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: SystImmune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-039-101
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioma; Solid Tumor
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): After the completion of the first cycle of treatment, if the patient has no intolerable toxic side effects during the first cycle of treatment, the investigator can communicate with the patient whether to continue the treatment during the 2-8 cycle.
  Interventions: Drug: GNC-039

INTERVENTIONS:
Drug: GNC-039 — Administration by intravenous infusion.

SUMMARY:
In this study, the safety, tolerability and preliminary effectiveness of GNC-039 in patients with relapsed/refractory or metastatic glioma or other solid tumors will be investigated to assess the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) or maximum administered dose (MAD) for MTD is not reached of GNC-039.

ELIGIBILITY:
Inclusion Criteria:

1. After failure of standard treatment (surgery, stupp regimen), subjects with diagnosed recurrent high-grade glioma (WHO Grade III-IV), or other recurrent/refractory or metastatic solid tumors can understand the informed consent, voluntarily participate in and sign the informed consent.
2. No gender limitation.
3. Age: ≥18 years old.
4. KPS≥60 points.
5. The expected survival as determined by the researchers was ≥3 months.
6. Hematological functions meet the following requirements: neutrophil absolute count (ANC) ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥90g/L.
7. Renal function meets the following requirements: creatinine (Cr) ≤1.5 ULN and creatinine clearance (Ccr) ≥50 mL/min (based on the calculation criteria of the study center), urinary protein ≤2+ or < 1000mg/24h (urine).
8. Liver functions meet the following requirements: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0×ULN; Total bilirubin ≤1.5×ULN (Gilbert's syndrome ≤3×ULN).
9. Coagulation function: fibrinogen ≥1.5g/L; Activated partial thromboplastin time (APTT) ≤1.5×ULN; Prothrombin time (PT) ≤1.5×ULN.
10. A fertile female subject or a fertile male subject with a fertile partner must use highly effective contraception from the date of informed consent until 12 weeks after the last dosing. Serum pregnancy tests must be negative for fertile female subjects within -10 to -3 days prior to initial dosing.
11. Subject is able and willing to comply with visits, treatment plans, laboratory tests, and other study-related procedures as specified in the study protocol.
12. For glioma patients: a. There must be a pathological diagnosis and a definite diagnosis of high-grade glioma; b. MRI diagnosis supported recurrence; c. Presence of at least one measurable tumor lesion according to RANO criteria; Or subjects receiving surgical treatment after recurrence; d. Archived primary or recurrent tumor tissue or sections that can be submitted to the Center for review (no less than 10 pathological white slices of 3-5μm or corresponding tissue blocks should be provided). If patients are unable to provide tumor tissue specimens, the Center may inform the sponsor and enroll them.
13. For patients with other solid tumors: a. Histologically or cytologically confirmed recurrent/refractory or metastatic solid tumors with disease progression confirmed by imaging or other objective evidence after standard treatment; Or subjects with refractory solid tumors who cannot tolerate standard therapy or have contraindications to standard therapy; b. Must have at least one measurable lesion that meets the RECIST v1.1 definition.

Exclusion Criteria:

1. Patients who are allergic to immunoglobulin or any component of the injectable formulation of GNC-039.
2. Patients with active infections requiring intravenous antibiotics who did not complete treatment 1 week prior to enrollment, except those who received prophylactic antibiotics for puncture or biopsy.
3. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBsAg positive or HBcAb positive with HBV-DNA copy number ≥ULN) or hepatitis C virus infection (HCV-RNA≥ULN).
4. Toxicity from prior antitumor therapy did not decrease to ≤ grade 1 as defined in CTCAE version 5.0 (except for toxicities that the investigators judged to be of no safety risk, such as alopecia, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy, etc.).
5. Patients at risk for active autoimmune diseases, or with a history of autoimmune diseases that may involve the central nervous system, Including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, Wegener syndrome, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. Exceptions include type I diabetes mellitus, hypothyroidism stable on hormone replacement therapy (including hypothyroidism caused by autoimmune thyroid disease), psoriasis or vitiligo that do not require systemic therapy, and autoimmune diseases caused by B cells and anti-autoimmune antibodies.
6. Lung disease defined by NCI-CTCAE v5.0 as ≥ grade 3, including patients with resting dyspnea, or in need of continuous oxygen therapy, or with a history of interstitial lung disease (ILD).
7. Previous organ transplant recipients.
8. History of severe cardiovascular and cerebrovascular diseases, including but not limited to: severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree III atrioventricular block, etc.; At rest, the QT interval was prolonged (QTc > 450 msec in men or 470 msec in women); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to initial administration; There is heart failure ≥II on the New York Heart Association (NYHA) cardiac function scale.
9. Thrombotic events such as deep vein thrombosis, arterial thrombosis, and pulmonary embolism occurred within 6 months prior to screening.
10. Other conditions deemed unsuitable for participation in this clinical trial by the investigator.
11. Brain gliomas: a. Patients who underwent surgery, chemotherapy, targeted and immunotherapy, iodine in vivo radiation, radiation therapy, or planned to undergo radiation therapy during the trial within 4 weeks of enrollment or 5 half-lives, whichever is shorter; b. Patients who had received intracranial lesion puncture biopsy within 7 days prior to enrollment; c. Received other investigational drugs or treatments that are not on the market within 4 weeks prior to enrollment; d. There was a history of central nervous system bleeding/infarction not associated with antineoplastic agents, such as stroke or intracranial and ocular bleeding (including embolic stroke), during the 6 months prior to enrollment.
12. For other solid tumors: a. Received chemotherapy, antibody therapy, molecular-targeted therapy, or investigational drugs within 4 weeks or 5 half-lives (whichever is shorter) of initial administration; b. Patients who underwent major surgery within 28 days prior to administration of the drug or were scheduled to undergo major surgery during the study period (except for procedures such as puncture or lymph node biopsy); c. poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg); d. Previous or associated central nervous system lesions, including but not limited to: paralysis, stroke (except those with lacunar infarction indicated by imaging examination but without treatment), severe brain injury, senile dementia, Parkinson's disease, organic brain syndrome, and psychosis; e. Received other investigational drugs or treatments that were not on the market within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 14 days after the first dose of GNC-039
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Maximum tolerated dose (MTD) or maximum administrated dose (MAD) | Up to 14 days after the first dose of GNC-039
  In the dose increment stage, the highest dose whose estimated DLT rate is closest to the target DLT rate but does not exceed the upper bound of the equivalent interval of DLT rate is selected as MTD.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  The incidence and severity of adverse events (TEAE) during treatment were graded according to the National Cancer Institute Standard for Common Terminology for Adverse Events (NCI-CTCAE, v5.0).

SECONDARY OUTCOMES:
Drug-related Adverse Events | Up to approximately 24 months
  Adverse Event (AE) refers to all adverse medical events that occur after a subject receives the investigational drug. Ae may be manifested as symptoms, signs, disease, or abnormalities in laboratory tests, but may not necessarily have a causal relationship with the investigational drug.
Cmax: Maximum serum concentration of GNC-039 | Up to 14 days after the first dose of GNC-039
  Maximum serum concentration (Cmax) of GNC-039 will be investigated.
Tmax: Time to maximum serum concentration (Tmax) of GNC-039 | Up to 14 days after the first dose of GNC-039
  Time to maximum serum concentration (Tmax) of GNC-039 will be investigated.
T1/2: Half-life of GNC-039 | Up to 14 days after the first dose of GNC-039
  Half-life (T1/2) of GNC-039 will be investigated.
AUC0-inf: Area under the serum concentration-time curve from time 0 to infinity | Up to 14 days after the first dose of GNC-039
  Blood concentration - Area under time line.
AUC0-t: Area under the serum concentration-time curve from time 0 to the time of the last measurable concentration | Up to 14 days after the first dose of GNC-039
  Blood concentration - Area under time line.
CL: Clearance in the serum of GNC-039 per unit of time | Up to 14 days after the first dose of GNC-039
  To study the serum clearance rate of GNC-039 per unit time.
Incidence and titer of ADA (Anti-drug antibody) | Up to approximately 24 months
  Frequency and titer of anti-GNC-039 antibody (ADA) will be evaluated.
ORR (Objective Response Rate ) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
OS (Overall Survival) | Up to approximately 24 months
  Overall survival is the time from randomization to death from any cause.
PFS (Progression-free Survival) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-039 to the first date of either disease progression or death, whichever occurs first.
DOR (Duration of Response) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Tiantan Hospital
Locations (6):
- China (6):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xian, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No